CLINICAL TRIAL: NCT06981585
Title: Comparison of Muscle Strength, Physical Activity, Sleep Quality and Quality of Life Between Children With Chronic Kidney Failure and Healthy Children
Brief Title: Physical Impairments in Children With Chronic Renal Failure
Status: Recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Principal Investigator, Izmir Democracy University
Other Study IDs: Healthy and Kidney Failure
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Failure; Chronic Kidney Diseases
Keywords: Chronic Kidney Failure; Muscle Strength; Physical Activity; Sleep Quality; Quality of Life
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Motor Activity; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Kidney Failure Group: This group will consist of children and adolescents with chronic kidney failure.
  Interventions: Other: Physical Evaluations of Patients with Chronic Kidney Failure
- Control Group: This group will consist of healthy children and adolescents.
  Interventions: Other: Physical Evaluations of Healthy Children

INTERVENTIONS:
Other: Physical Evaluations of Patients with Chronic Kidney Failure — In this study, data from children and adolescents with chronic kidney disease will be collected through face-to-face assessments. Grip strength, cough strength, physical activity, sleep quality and quality of life will be assessed in children and adolescents who meet the inclusion criteria. All data obtained through these assessments will be collected from participants face-to-face at one time and for a maximum of approximately 1 hour.
  Groups: Chronic Kidney Failure Group
Other: Physical Evaluations of Healthy Children — In this study, data from healthy children and adolescents will be collected through face-to-face assessments. Grip strength, cough strength, physical activity, sleep quality and quality of life will be assessed in children and adolescents who meet the inclusion criteria. Data obtained through all these assessments will be collected from participants face-to-face at once and for a maximum of approximately 1 hour.
  Groups: Control Group

SUMMARY:
When the literature is examined, it is seen that the extent to which cough strength, grip strength, physical activity level and quality of life levels are affected in children with chronic kidney failure compared to healthy children is not sufficiently clarified. For this reason, this study aimed to reveal impairments in grip strength, cough strength, physical activity, sleep quality or quality of life in children with chronic renal failure compared to healthy children.

DETAILED DESCRIPTION:
The aim of this study is to compare children and adolescents with chronic kidney disease with healthy children and adolescents in terms of grip strength, cough strength, physical activity, sleep quality and quality of life. Participants will be evaluated for these parameters through clinical assessments, questionnaires and measurements. The aim of the study is to understand the health effects of chronic kidney disease and to provide the basis for improvements in the health management of these individuals.

ELIGIBILITY:
Inclusion Criteria: for Children and Adolescents with Chronic Kidney Failure

* Being between the ages of 8-18
* Being clinically stable for at least the last 3 weeks
* Having the necessary cooperation for the measurements
* Being willing to participate in the study

Inclusion Criteria for Healthy Children and Adolescents:

* Being between the ages of 8-18,
* Having the necessary cooperation for the measurements,
* Being willing to participate in the research

Exclusion Criteria: for Children and Adolescents with Chronic Kidney Failure

* Having any orthopedic, neurological, cardiovascular or psychological problems that may prevent measurements from being taken in the last 6 months
* Being a smoker or having quit
* Having had a kidney transplant.

Exclusion Criteria for Healthy Children and Adolescents:

* Having a history of any orthopedic, neurological, cardiovascular or psychological problems that may prevent measurements from being taken in the last 6 months
* Having any chronic disease
* Being a smoker or having quit smoking

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: At least 25 patients with Chronic Kidney Failure will be included in the research group and at least 25 healthy individuals will be included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life score | through study completion, an average of 1 year
  The scale we will use to assess health-related quality of life, the Pediatric Quality of Life Inventory (PedsQL 4.0). The scale was developed to assess the health-related quality of life of children and adolescents between the ages of 2 and 18 and consists of physical, emotional, social and school functioning items, totaling 23 items.Scores from this questionnaire are converted to a scale of 0 to 100. Higher scores indicate better health-related quality of life.

SECONDARY OUTCOMES:
Cough Strength | through study completion, an average of 1 year
  The peak cough expiratory flow (PEF) of the individual will be assessed in the upright sitting position using a peak cough flow meter (PEF meter) (Expirite Peak Flow Meter, China). The individual coughs into the PEF meter as forcefully as possible following deep inspiration. The best of at least three repetitions is recorded.
Hand Grip Strength | through study completion, an average of 1 year
  Grip strength will be measured using a dynamometer. Each hand will be tested three times, and the highest value will be recorded for both sides.
Evaluation of Physical Activities | through study completion, an average of 1 year
  The Godin-Shephard leisure-time physical activity questionnaire will be used to determine the number of times individuals engage in physical activity during a one-week period. The questionnaireasks how many times individuals engage in physical activity lasting at least 15 minutes or longer during their free time over a 7-day period. This is used to calculate individuals' total physical activity scores. The higher the total score, the higher the individual's physical activity level. According to the score obtained from this questionnaire using moderate and strenuous physical activities; those who score 24 units or more are classified as Active (Significant benefits), those who score between 14-23 units are classified as Moderately active (Some benefits), and those who score less than 14 units are classified as Insufficiently active (Less important or low benefits).
Evaluation of sleep quality | through study completion, an average of 1 year
  Children's Sleep Habits Questionnaire-Short Form will be used to evaluate sleep disorder in individuals and it consists of a total of 33 items.The total score is calculated.The lowest possible score for the questionnaire is 0, and the highest is 99. The higher the total score, the more sleep problems the individual has.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Barğı, Study Director — İzmir Demokrasi Üniversitesi; Hüseyin Kıran, Principal Investigator — İzmir Demokrasi Üniversitesi; Nida Dinçel, Study Director — SBÜ İTF DR. BEHÇET UZ ÇOCUK HASTALIKLARI VE CERRAHİSİ EĞİTİM VE ARAŞTIRMA HASTANESİ
Locations (1):
- İzmir Demokrasi Üniversitesi, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clark SL, Denburg MR, Furth SL. Physical activity and screen time in adolescents in the chronic kidney disease in children (CKiD) cohort. Pediatr Nephrol. 2016 May;31(5):801-8. doi: 10.1007/s00467-015-3287-z. Epub 2015 Dec 18. PMID 26684326
- [Background] Taner S, Ekberli G, Gunes S. The Effect of Sleep Habits on Quality of Life in Pediatric Patients With Chronic Kidney Disease. Cureus. 2024 Jul 15;16(7):e64585. doi: 10.7759/cureus.64585. eCollection 2024 Jul. PMID 39144881
- [Background] Darwish AH, Abdel-Nabi H. Sleep disorders in children with chronic kidney disease. Int J Pediatr Adolesc Med. 2016 Sep;3(3):112-118. doi: 10.1016/j.ijpam.2016.06.001. Epub 2016 Jun 29. PMID 30805480